CLINICAL TRIAL: NCT07123051
Title: Robotic Assisted Right Colectomy With the DEXTER Robotic Surgery System
Acronym: RACER
Status: Recruiting | Type: Observational
Sponsor: Distalmotion SA (Industry)
Collaborators: Confinis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-01
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Right Colectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: right colectomy — Robotic-assisted right colectomy with the DEXTER robotic surgery system

SUMMARY:
This study aims to confirm the perioperative and early postoperative safety and clinical performance (efficacy) of the Dexter Robotic System, in patients undergoing robotic-assisted right colectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Patient agrees to perform the 30-day follow-up assessment as per standard of care

Exclusion Criteria:

* History of radiotherapy on the target surgical area
* Patients with distant metastasis
* Any planned concomitant procedures
* History of major abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing a right colectomy for malignant or benign indication
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary safety outcome | up to 30 days after surgery
  Occurrence of Clavien-Dindo grades III-V adverse events
Primary efficacy outcome | Intraoperative
  Successful completion of the Dexter-assisted procedure, i.e. free of any device related conversion to an open or fully laparoscopic surgical approach.

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - CH Châteauroux - Le Blanc, Châteauroux
  - Groupe Hospitalier Saintes - Saint-Jean-d'Angély, Saintes, Saintes
- Artemed Klinikum München Süd, Munich, Germany